CLINICAL TRIAL: NCT06527391
Title: Supplemental Choline to Prevent and Treat Learning and Memory Deficits of Early Iron Deficiency: the SupCHO Study
Brief Title: Choline and Iron Deficiency
Status: Recruiting | Phase: Phase 2 / Phase 3 | Type: Interventional
Sponsor: University of Minnesota (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Prevention
Other Study IDs: 33410
Record Dates: First submitted 2024-07-24; First posted 2024-07-30 (Actual); Last update posted 2025-08-27 (Actual); Status verified 2025-08

CONDITIONS: Pediatric Iron Deficiency; Anemia
Keywords: iron deficiency; choline; anemia
MeSH Terms: conditions — Anemia; Iron Deficiencies | interventions — Choline

STUDY DESIGN:
Intervention Model Description: Randomized, double-blinded, placebo-controlled trial of 9 months of daily choline supplementation of 300 6-month-old Ugandan infants with iron deficiency anemia
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: Manufacturer of choline and placebo tablets will randomize the regimens and hold the randomization key
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- study group (Experimental): participants assigned to receive study drug
  Interventions: Drug: choline bitartrate
- control group (Placebo Comparator): participants assigned to receive placebo drug
  Interventions: Other: placebo drug

INTERVENTIONS:
Drug: choline bitartrate — Daily supplementation for 9 months with 200 mg choline bitartrate
  Arms: study group
Other: placebo drug — Daily supplementation for 9 months with identical placebo
  Arms: control group

SUMMARY:
BACKGROUND:

Iron deficiency limits the neurodevelopmental potential of more than 200 million children each year. Iron therapy is typically started when iron deficiency anemia is first diagnosed after screening for anemia or detection of clinical symptoms of iron deficiency anemia at 12 months of age. But iron started at this time does not fully correct earlier iron-deficiency-mediated brain dysfunction, underscoring the need for low-cost, easily implementable adjunct therapies to iron to treat or prevent this dysfunction in high-risk populations.

GAP Supplementation with the nutrient choline lessens damage to the hippocampus from early-life iron deficiency in pre-clinical models and improves hippocampus-mediated memory in children with Fetal Alcohol Spectrum Disorders. Choline has not been tested in children with iron deficiency anemia, despite strong pre-clinical and clinical evidence supporting a benefit to brain development.

HYPOTHESIS:

Infants with iron deficiency anemia who receive iron and nine months of daily choline supplements will have better scores on specific neurobehavioral tests of recognition memory than infants who receive iron and placebo.

METHODS:

This randomized, double-blinded, placebo-controlled clinical trial will randomize 300 6-month-old infants with iron deficiency anemia at Mulago Hospital, Kampala, Uganda, to iron plus choline or iron plus placebo to test the effect of choline on hippocampus-specific and global neurobehavioral outcomes after nine months.

RESULTS: Pending

IMPACT:

If our hypothesis is correct, choline could be added immediately to standard-of-care treatment for iron deficiency anemia. This intervention could safely mitigate the brain dysfunction of early-life iron deficiency that is often undiagnosed until the hippocampal critical window is closing. This simple, low-cost nutrient could thus have life-long benefit for both individuals and the economic and social prosperity of entire regions.

ELIGIBILITY:
Inclusion Criteria:

* Age 6 months +/- 28 days
* Hb < 11.0 g/dL
* ZPP > = 80
* T<37.5°C
* Malaria-negative based on Rapid Diagnostic Test (RDT)
* Mother is HIV-negative.

Exclusion Criteria:

* Developmental disorder
* Severe malnutrition (severe wasting or bipedal edema)
* Known sickle cell disease
* Neurologic disorder, brain injury, or other condition affecting brain development
* Not currently breastfeeding
* Birthweight < 2000 g

Ages: 5 Months to 7 Months | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 300 (Estimated)
Dates: Start 2025-08-11 (Actual); Primary Completion 2027-09-21 (Estimated); Study Completion 2027-09-21 (Estimated)

PRIMARY OUTCOMES:
Elicited Imitation score | 9 months (1 month = 28 days) after enrollment
  Elicited Imitation outcomes (number of items correctly recalled and number of steps recalled in the correct order for both immediate and delayed recall) at age 15 months, i.e., after nine months of daily supplementation with choline or placebo.
1) Composite Score on the Mullen Scales of Early Learning; 2) Behavior Rating Scale (BRS) composite score; 3) Early Childhood Vigilance Test (ECVT, computerized test for attention). | 9 months (1 month = 28 days) after enrollment
  1) Composite Score on the Mullen Scales of Early Learning; 2) Behavior Rating Scale (BRS) composite score; 3) Early Childhood Vigilance Test (ECVT, computerized test for attention).

CONTACTS AND LOCATIONS:
Overall Officials: Sarah Cusick, Principal Investigator — University of Minnesota
Locations (1):
- University of Minnesota, Minneapolis, Minnesota, United States

REFERENCES:
- [Derived] Cusick SE, Mupere E, Bangirana P, Baluku RI, Kroupina M, Cheatham CL, Wozniak JR, Georgieff MK. Supplemental choline to prevent and treat learning and memory deficits of early-life iron deficiency (The SupCHO Study): study protocol for a randomized, placebo-controlled trial in Ugandan infants with iron deficiency anemia. Trials. 2025 Nov 19;26(1):524. doi: 10.1186/s13063-025-09246-2. PMID 41257751